CLINICAL TRIAL: NCT05037292
Title: PAtient-centered mUltidiSciplinary Care for vEterans Undergoing Surgery (PAUSE): a Hybrid 1 Clinical Effectiveness-implementation Intervention Trial
Brief Title: PAtient-centered mUltidiSciplinary Care for vEterans Undergoing Surgery (PAUSE)
Acronym: PAUSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 20-077; 1I01HX003215-01A1 (NIH)
Record Dates: First submitted 2021-08-10; First posted 2021-09-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Frailty
Keywords: Surgery; Multidisciplinary care model; Implementation science; Pragmatic clinical trial; Qualitative research; Randomized Controlled Trial
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Onboarding, training, and implementation of surgical subspecialties into a standardized frailty screening index and the utilization of a frailty review board by surgical specialty.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PAUSE (Experimental): Surgical specialty clinics that completed an "onboarding" training for team members to use the standardized frailty screening incorporated in Veterans' medical records. Veterans identified as frail upon screening will be referred to a multidisciplinary "PAUSE Board" comprised of members from surgery, anesthesia, geriatrics, palliative care, case management, rehabilitation, nutrition.
  Interventions: Other: PAUSE Intervention
- Usual Care (No Intervention): Surgical specialty clinics that have not yet implemented the PAUSE Intervention. Veterans at these clinics will receive usual perioperative assessment and management by the clinical team.

INTERVENTIONS:
Other: PAUSE Intervention — Standardized frailty screening and utilization of a frailty review board (PAUSE Board)
  Other Names: frailty screening; utilization of frailty review board
  Arms: PAUSE

SUMMARY:
The PAUSE Trial is a pragmatic, randomized clinical trial for Veterans scheduled for elective surgery at 3 large VA facilities (Palo Alto, Houston, and Nashville). The PAUSE Trial focuses on cooperation between providers of various disciplines in order to provide better care. Veterans identified as frail upon standardized will be referred to a multidisciplinary "PAUSE Board" comprised of members from surgery, anesthesia, geriatrics, palliative care, case management, rehabilitation, and nutrition. Diverse specialists will come together in a team environment to discuss care options, scientific evidence, and patient goals and expectations, creating individual patient recommendations. The investigators hypothesize that the PAUSE Board model will improve quality and outcomes by promoting guidelines and evidence-based care recommendations as well as constructive team-based discussions to align care with patient goals and expectations.

DETAILED DESCRIPTION:
Background: Frailty is a syndrome of reduced physiologic reserve associated with higher postoperative mortality and adverse outcomes. The investigators' preliminary work shows that institution-wide frailty screening and introducing a "pre-surgical pause" reduces 6-month mortality threefold. However, a knowledge gap exists in the nature of the intervention and which stakeholders should be involved in the "pre-surgical pause". Multidisciplinary care models for complex patients are highly effective in oncology, wound care and primary care. The investigators propose a new care delivery model, i.e. PAtient-centered mUltidiSciplinary care for vEterans undergoing surgery (PAUSE), where experts from diverse fields contribute to surgical decision-making and optimize outcomes for high-risk Veterans.

Impact: Veterans above 65 years-of-age are a fast-growing population with significant need for high-quality surgical care. This study builds a structured multidisciplinary workflow to improve clinical and quality outcomes and provides high-value care for frail and high-risk Veterans that aligns with VA priorities and patient goals and expectations.

Innovation: This is the first study in the VA to implement a multidisciplinary care model for surgical care. The intervention employs an innovative hybrid-1 clinical effectiveness-implementation design to evaluate novel Veteran-centric outcomes of 30- and 180-day mortality, non-home discharge, rehospitalizations and home-time. A detailed formative evaluation (FE) evaluates provider and system factors that impact PAUSE intervention uptake. Further, the study has support from three national operational partners: National Surgery Office, Office of Geriatrics and Extended Care, and Palliative Care and Hospice Program.

Specific Aims: The goals for this project are to: (1) test the effectiveness of the PAUSE trial intervention vs usual care in improving 30- and 180-day mortality, non-home discharge, rehospitalizations and home-time for patients undergoing surgical evaluation; (2) test moderators of the PAUSE intervention effectiveness (treatment effect heterogeneity), especially specialty, frailty severity and risk status; and (3) use a mixed-method FE to understand the factors that influence fidelity, adaptation, and implementation of the PAUSE intervention. The investigators hypothesize that the PAUSE intervention will decrease 30- and 180-day mortality, rehospitalizations, and non-home discharge and increase home-time for all Veterans (Aim 1). The effect size for the outcomes will be greater for frail patients in certain specialties (Aim 2). The concurrent FE will highlight key barriers/facilitators for future implementation (Aim 3).

Methodology: The PAUSE trial is a pragmatic, stepped-wedge randomized clinical trial designed to capture a cohort of 25,000 Veterans scheduled for elective surgery at 3 large tertiary care VAMCs (Palo Alto, Houston and Nashville) and 7 specialty groups in each center: general, vascular, orthopedics, cardio-thoracic, urology, neurosurgery and others (e.g., plastics and ENT). The intervention includes standardized frailty screening and referral to a "multidisciplinary PAUSE Board" (surgery, anesthesia, geriatrics, palliative care, case management, rehabilitation and nutrition) for recommendations. Each 'step' is a randomly chosen specialty transitioning from usual care to the PAUSE intervention. Outcomes include 30- and 180-day mortality, non-home discharge, rehospitalizations and home-time. The Consolidated Framework for Implementation Research is used to guide FE and analysis of factors that influence implementation. The study spans across 4-years for pre-intervention FE (Y1), PAUSE intervention (Y1-3), post-intervention FE (Y3) and analysis (Y4).

ELIGIBILITY:
Inclusion Criteria:

Chart/Database Review:

* Patient must have elective surgery within the intervention period
* Surgery must be with a qualifying specialty (general, vascular, orthopedics, cardio-thoracic, urology, neurosurgery, and others [e.g., Plastics/ENT])
* Surgery must be at either the VA Palo Alto, VA Houston, or VA Nashville

VA Providers:

* Service and Section Chief Interviews:

  * Must be the Surgery Service Line chief (or appointed designee).
  * Must be Section Chief (or appointed designee) of a qualifying surgical specialty (general, vascular, orthopedics, cardio-thoracic, urology, neurosurgery, and others [e.g., Plastics/ENT]).
  * Must serve at the VA Palo Alto, VA Houston, or VA Nashville.
* Focus Groups:

  * Must be a healthcare provider at VA Palo Alto, VA Houston, or VA Nashville.
  * Must have planned or prior experience participating in PAUSE Board meetings.
* Referral Frequency Interviews:

  * Must be a member of the surgical team with one of the qualifying surgical specialties (general, vascular, orthopedics, cardio-thoracic, urology, neurosurgery, and others [e.g., Plastics/ENT]).
  * Must be one of the high- or low-referring providers to the PAUSE Board.

Exclusion Criteria:

Chart/Database Review:

-Non-Veteran (USA)

VA Providers:

-Refusal or inability to participate during site visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35015 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
180-day mortality | Up to 180-days after discharge
  The rate of mortality at or within 180 days after the elective surgery

SECONDARY OUTCOMES:
30-day mortality | Up to 30-days after discharge
  The rate of mortality at or within 30 days after the elective surgery
30-day rehospitalization | Up to 30-days after discharge
  The percent of rehospitalizations at or within 30 days after the elective surgery
180-day rehospitalization | Up to 180-days after discharge
  The percent of rehospitalizations at or within 180 days after the elective surgery
Non-home discharge | 1 day after surgery discharge
  The percent of non-home discharge dispositions
180-day home-time | Up to 180-days after discharge
  The percent of time spent at home (vs. non-home environment) in the 180 days after elective surgery

OTHER OUTCOMES:
Risk Analysis Index | Up to 90 days before surgery
  Frailty assessment where higher scores indicates higher frailty [0=lowest frailty, 81=highest frailty].
Care Assessment Need | Up to 90 days before surgery
  A predictive analytic tool for hospitalization and death at 90 days and one year, generated from electronic health records to assist Patient Aligned Care Teams in patient management and care coordination. Percentile score calculated where higher percentile indicates higher risk [0=lowest risk, 99=highest risk].
Operative Stress Score | Through study completion, an average of 1 year
  Score indicates the physiological stress of a surgery using CPT codes in the electronic health records [1=very low stress, 5=very high stress].
Activities of Daily Living--long form | Through study completion, an average of 1 year
  Total score reflects an individual's ability to complete basic self-care activities independently on 7 items (e.g., locomotion, eating) [0=completely independent, 28=completely dependent].
Activities of Daily Living--short form | Through study completion, an average of 1 year
  Total score reflects an individual's ability to complete basic self-care activities independently on 4 items (e.g., locomotion, ) [0=completely independent, 16=completely dependent].
Instrumental Activities of Daily Living--Difficulty Scale | Through study completion, an average of 1 year
  Total score reflects an individual's ability to accomplish tasks needed for self-maintenance and independence on 3 items [0=independent, 6=dependent].
Instrumental Activities of Daily Living--Involvement Scale | Through study completion, an average of 1 year
  Score reflects an individual's ability to accomplish tasks needed for self-maintenance and independence on 3 items [0=independent, 21=dependent].
Survey of Healthcare Experiences of Patients Care Coordination | Through study completion, an average of 1 year
  Percent of "Always" (4=Always) responses where scores on 3 items reflect satisfaction with care coordination; each item 1=Never, 2=Sometimes, 3=Usually, 4=Always. Higher percent indicates better care coordination.
Survey of Healthcare Experiences of Patients Care Transition | Through study completion, an average of 1 year
  Percent of "Strongly Agree" responses where scores on 3 items reflect satisfaction with care coordination; each item 1=Strongly Disagree, 2=Disagree, 3=Agree, 4=Strongly Agree. Higher percent indicates better care transition.
Survey of Healthcare Experiences of Patients--Inpatient | Through study completion, an average of 1 year
  Facility level scores of patient satisfaction with hospitalization where higher scores indicate higher patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Shipra Arya, MD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT05037292/ICF_000.pdf